CLINICAL TRIAL: NCT04547829
Title: Safety and Efficacy of Pegylated Recombinant Human Granulocyte-colony Stimulating Factor(PEG-rhG-CSF) in Preventing Neutropenia in Children With Tumor After Chemotherapy：A Multi-center, Single Arm Trial.
Brief Title: Safety and Efficacy of PEG-rhG-CSF in Preventing Neutropenia in Children With Tumor After Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEG-rhG-CSF
Record Dates: First submitted 2020-09-11; First posted 2020-09-14 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEG-rhG-CSF (Experimental): pegylated recombinant human granulocyte-colony stimulating factor subcutaneous injection
  Interventions: Drug: pegylated recombinant human granulocyte-colony stimulating factor

INTERVENTIONS:
Drug: pegylated recombinant human granulocyte-colony stimulating factor — The dosage was determined according to the patient's weight, 100 UG / kg each time; The method of administration: subcutaneous injection; The time of administration: 24-48 hours after the end of chemotherapy, once in each chemotherapy cycle.

SUMMARY:
The purpose is to evaluate the safety of PEG-rhG-CSF in the prevention of neutropenia in children with tumor after chemotherapy, and then evaluate the effectiveness of PEG-rhG-CSF in preventing neutropenia in children with tumor after chemotherapy.

DETAILED DESCRIPTION:
The dosage was determined according to the patient's weight, 100 UG / kg each time; The method of administration: subcutaneous injection; The time of administration: 24-48 hours after the end of chemotherapy, once in each chemotherapy cycle.

ELIGIBILITY:
Inclusion Criteria:

- 1)6 years < age < 18 years old, regardless of gender; 2)Tumor patients diagnosed by histopathology or bone marrow cytology; 3)Patients who have not been treated for the first time; 4)ECoG score ≤ 2; 5)The expected survival time is more than 8 months; 6)The hematopoietic function of bone marrow was normal (ANC ≥ 1.5 × 109 / L, PLT ≥ 80 × 109 / L, Hb ≥ 75 g / L, WBC ≥ 3.0 × 109 / L); 7)Receive high-intensity chemotherapy, such as scccg lymphoma, CAV / ie, VIP regimen, etc., and expect bone marrow suppression of grade III or above after chemotherapy.

8)Patient's parent or guardian signs informed consent.

Exclusion Criteria:

* Patients with any of the following items will not be enrolled in this study:

  1. Local or systemic infection without adequate control;
  2. Severe visceral dysfunction;
  3. Liver function test: total bilirubin (TBIL), alanine aminotransferase (ALT), aspartate aminotransferase (AST) were all higher than 2.5 times of the upper limit of normal value; if due to liver metastasis, the above indicators were more than 5 times of the upper limit of normal value; renal function test: Serum creatinine (CR) > 2 times of the upper limit of normal value;
  4. Those who took the same kind of other tested drugs or accepted clinical trials of other drugs within 4 weeks before enrollment;
  5. Allergic to peg-rhG-CSF, rhG-CSF and other preparations or proteins expressed by Escherichia coli;
  6. Serious mental illness, affecting informed consent and / or expression or observation of adverse reactions;
  7. The researcher judged the patients who were not suitable to participate.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-10-10 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
safety of PEG-rhG-CSF in the prevention of neutropenia in children with tumor after chemotherapy | From the beginning of observation to the end of observation（6 weeks) of the last enrolled patient
  The incidence and severity of adverse events;

SECONDARY OUTCOMES:
To evaluate the effectiveness of PEG-rhG-CSF in preventing neutropenia in children with tumor after chemotherapy. | From the beginning of observation to the end of observation（6 weeks) of the last enrolled patient
  The incidence of grade III / IV ANC reduction in each chemotherapy cycle

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University CancerCenter
Locations (1):
- Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang J, Lu S, Wang J, Jiang L, Luo X, He X, Wu Y, Wang Y, Zhu X, Chen J, Tang Y, Chen K, Tian X, Shi B, Guo L, Zhu J, Sun F, Zhen Z, Zhang Y. A multicenter phase II trial of primary prophylactic PEG-rhG-CSF in pediatric patients with solid tumors and non-Hodgkin lymphoma after chemotherapy: An interim analysis. Cancer Med. 2023 Jul;12(13):14130-14137. doi: 10.1002/cam4.6079. Epub 2023 May 15. PMID 37183837